CLINICAL TRIAL: NCT05848557
Title: mSaada: A Mobile Health Tool to Improve Cervical Cancer Screening in Western Kenya
Brief Title: mSaada: A Mobile Health Tool
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Pro00108937
Record Dates: First submitted 2023-04-14; First posted 2023-05-08 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Cervical Cancer; HPV; mHealth
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Counseling will be provided using standard Ministry of Health (MoH) items and screening data and specimen tracking will be done using MoH registers.
- mSaada platform (Experimental): Counseling, specimen tracking and case management will be facilitated using mSaada.
  Interventions: Behavioral: mSaada

INTERVENTIONS:
Behavioral: mSaada — mSaada is an integrated digital platform to support patients, community health volunteers (CHVs), providers and health systems in an HPV-based cervical cancer screening strategy. mSaada is hosted on an open-source platform (Dimagi, CommCare) as a mobile health application to support patient data collection, protocol support and counseling aids. mSaada will include an education module, patient and specimen tracking, screening reminders, and messaging functionality.
  Arms: mSaada platform

SUMMARY:
In the R21 phase of this project, investigators will: (1) work with key stakeholders and local and international developers to finalize the mSaada platform, building on the existing prototype to add patient and specimen tracking functionality; and (2) carry out a pilot to identify the patient, provider and health system factors necessary to design a trial to evaluate mSaada effectiveness in assisting community health volunteer-led home-based HPV screening, and implementation factors. Investigators will carry out a six-month pilot of mSaada with community units in two health facilities providing HPV-based screening, and use performance metrics including system usage rates, workflow observations and qualitative data to guide the planning of a to determine effectiveness.

In the R33 phase of the project, investigators plan to: (1) conduct an 18-month c-RCT across 12 health facilities to determine the impact of mSaada on cervical cancer screening uptake, treatment acquisition and cervical cancer knowledge levels among women in the community; and (2) measure the requisite implementation factors for mSaada effectiveness, sustainability, and scale-up. The rigorous study design will allow us to determine the clinical impact of mSaada, ensure the local and regional infrastructure has the capacity necessary for sustainability and develop strategies for widespread implementation and scale-up. Collaboration with key stakeholders from the Kenya Ministry of Health will facilitate the development of a long-term sustainability plan as the country moves toward HPV-based cervical cancer screening. Investigators anticipate the mSaada platform will play a pivotal role in facilitating the introduction of HPV-based screening programs that can reach women in settings with limited health care infrastructure.

ELIGIBILITY:
R21

Aim 1 Community health volunteers (CHVs), facility providers and supervisors, Ministry of Health officials

Inclusion Criteria:

* 18 years or older
* be employed by a government clinic
* be working in cervical cancer screening

Exclusion Criteria:

* Does not understand the study purpose and details
* Is not willing to provide informed consent

Women

Inclusion Criteria:

- between 30 and 65 years old

Exclusion Criteria:

* Does not understand the study purpose and details
* Is not willing to provide informed consent

Aim 2 Community health volunteers (CHVs)

Inclusion Criteria:

* 18 years or older
* be employed by a government clinic
* be working in cervical cancer screening

Exclusion Criteria:

* Does not understand the study purpose and details
* Is not willing to provide informed consent

Women

Inclusion Criteria:

* between 30 and 65 years old
* intact cervix and uterus
* able to provide informed consent.

Exclusion Criteria:

* Does not understand the study purpose and details
* Is not willing to provide informed consent

R33

Women (knowledge and risk perception surveys) We plan to enroll approximately 600 women (50 per health facility) to complete a survey about cervical cancer and HPV knowledge, risk perception and screening awareness, acceptability and self-efficacy.\

Eligibility criteria for women participants include:

* Reside within Siaya County, in one of the study communities
* Eligible for cervical cancer screening per the Kenya Ministry of Health guidelines and
* Ability to provide informed consent.

CHPs in both arms will be asked to complete a survey about their self-efficacy, knowledge of HPV and cervical cancer, and the usability of the mSaada app (CHPs in the intervention arm only).

Inclusion:

* CHV participants must be employed by government clinics in Siaya County, and
* be able to provide informed consent.

Exclusion:

* Does not understand the study purpose and details
* Is not willing to sign an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Community Health Volunteers (CHVs) reporting a usability score greater than 60 | 1-day
  mSaada Usability Survey with a range of 20-100, where a higher score indicates a higher level of acceptability (mean scores >60 is considered acceptable).
Proportion of women in each arm who complete cervical cancer screening | 1-day
  Calculated by dividing the number of women screened by the number of eligible women attending health facilities
Proportion of women in each arm who test HPV-positive and access treatment within 3 months of receiving their results | 1-day
  Calculated the number of women treated within 3 months of receiving their results by dividing the number of women who test HPV positive
Difference in women's knowledge level of cervical cancer as measured by a knowledge scale between the arms | 1-day
  The knowledge scale has a score range of 0 to 5, where a higher score indicates a higher level of knowledge.
Difference in women risk perception of cervical cancer as measured by a risk perception scale between the arms | 1-day
  The Risk Perception Scale has 3 Likert scale questions regarding risk perception.
Difference in Community Health Promoter (CHP) screening self-efficacy, knowledge, usability between the arms | 1-day
  Quantitative self-efficacy, knowledge and usability survey with CHPs after participating in the study..

CONTACTS AND LOCATIONS:
Locations (1):
- Kenya Medical Research Institute, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF